CLINICAL TRIAL: NCT04120298
Title: Effects of Structured and Individualized Exercise in Patients With Metastatic Breast Cancer on Fatigue and Quality of Life
Brief Title: Effects of Exercise in Patients With Metastatic Breast Cancer
Acronym: EFFECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: German Cancer Research Center (Other); Australian Catholic University (Other); Karolinska Institutet (Other); The Netherlands Cancer Institute (Other); Medical University of Gdansk (Other); Fundación Onkologikoa Fundazioa (Unknown); Europa Donna (Unknown); German Sport University, Cologne (Other); University Hospital Heidelberg (Other); Nurogames GmbH, Cologne (Unknown)
Responsible Party: Principal Investigator, Dr. Anne May, Cancer Epidemiologist, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-524; NL69600.041.19 (Other: CCMO)
Record Dates: First submitted 2019-09-12; First posted 2019-10-09 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Breast Cancer
Keywords: exercise; cancer-related fatigue; quality of life
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised exercise group (Experimental): The intervention group will participate in a 9-month exercise intervention. The exercise program will start with a 6-month period, where patients participate in a supervised multimodal exercise program twice a week supplemented with unsupervised exercises. The multimodal exercise program comprises aerobic-, resistance- and balance components. After completing the initial six-month period, one supervised session will be replaced by one unsupervised session until month nine.
  Unsupervised exercises will be supported by an activity tracker (FitBit) and an exercise App specifically designed for the EFFECT trial
  Interventions: Behavioral: Supervised exercise
- Control group (No Intervention): Patients randomized to the control group will also receive an activity tracker (like the intervention group). We will advice control patients to avoid inactivity and be as physically active as current abilities and conditions allow, with the aim to progress towards being physically active for 150min/week in line with the current exercise guidelines.

INTERVENTIONS:
Behavioral: Supervised exercise — An individualised exercise programme supervised by a trained instructor
  Arms: Supervised exercise group

SUMMARY:
Currently, the effect of exercise on metastatic breast cancer has not been extensively studied, even though the benefits are evident in the curative setting. The investigators designed the EFFECT study to assess the effects of a 9-month structured and individualised exercise intervention in 350 patients with metastatic breast cancer (stage IV) on cancer-related physical fatigue, Health-Related Quality of Life (HRQoL), and other disease and treatment-related side effects at six months (primary endpoint).

DETAILED DESCRIPTION:
The EFFECT study is a multicentre, randomised controlled trial. The intervention group will participate in a 9-month exercise intervention. The exercise program will start with a 6-month period, where patients participate in a supervised multimodal exercise program twice a week supplemented with unsupervised exercises. The multimodal exercise program comprises aerobic-, resistance- and balance components. After completing the initial six-month period, one supervised session will be replaced by one unsupervised session until month nine.

Unsupervised exercises will be supported by an activity tracker (FitBit) and an exercise App specifically designed for the EFFECT trial. Patients randomized to the control group will also receive an activity tracker (like the intervention group). The investigators will advice control patients to avoid inactivity and be as physically active as current abilities and conditions allow, with the aim to progress towards being physically active for 150min/week in line with the current exercise guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer stage IV
* ECOG (Eastern Cooperative Oncology Group scale) performance status ≤ 2
* Able and willing to perform the exercise program and wear the activity tracker

Exclusion Criteria:

* A potential subject who meets any of the following criteria is not eligible for enrolment into this study:

  * Unstable bone metastases inducing skeletal fragility as determined by the treating clinician
  * Untreated symptomatic known brain metastasis
  * Estimated life expectancy < 6 months as determined by the treating clinician
  * Serious active infection
  * Too physically active (i.e. >210 minutes/week of moderate-to-vigorous intentional exercise
  * Severe neurologic or cardiac impairment according ACSM criteria
  * Uncontrolled severe respiratory insufficiency as determined by the treating clinician or if the patient is dependent on oxygen suppletion in rest or during exercise
  * Uncontrolled severe pain
  * Any other contraindications for exercise as determined by the treating physician
  * Any circumstances that would impede adherence to study requirements or ability to give informed consent, as determined by the treating clinician
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Cancer-related physical fatigue | 0- 6 months (measured at baseline, 3 and 6 months)
  Physical fatigue measured with the EORTC QLQ-FA12
Health-related Quality of Life | 0- 6 months (measured at baseline, 3 and 6 months)
  Disease specific HRQoL measured with the EORTC QLQ-C30 Summary Score

SECONDARY OUTCOMES:
Separate HRQoL domains and Summary Score | 0-9 months
  EORTC QLQ-C30 function and symptom scores scores
Cancer-related fatigue | 0-9 months
  EORTC QLQ-FA12 scores
Breast cancer specific symptoms | 0-9 months
  EORTC QLQ-BR45
Anxiety, depression | 0-9 months
  PHQ-4
Sleep | 0-9 months
  PSQI
Pain: severity and its impact on functioning. | 0-9 months
  BPI
Neuropathic pain | 0-9 months
  painDETECT
Pain Catastrophizing | 0-9 months
  PCS
Treatment-related toxicities grade≥3 | 0-9 months
  Common Toxicity Criteria for adverse events (CTCAE)
Weight | 0-6 months
  weight measured in KG
Height | 0-6 months
  Height measured in meters
Waist circumference | 0-6 months
  waist circumference measured in cm
Body composition (fat free mass and fat mass) | 0-6 months
  Bioelectrical impedance analysis (BIA), add-on in some centers (not obligatory): DEXA
Physical activity (subjective) | 0-6-9 months
  Questionnaire
Physical activity (objective) | 0-6-9 months
  activity tracker
Resting heart rate | 0-6 months
  Resting heart rate
Blood pressure | 0-6 months
  Blood pressure (diastolic and systolic) measured at rest
Physical performance | 0-6 months
  Short Physical Performance Battery, handgrip- and leg strength test
Physical fitness | 0-6 months
  Steep ramp test and endurance cycle test, add-on (not obligatory): CPET
Work status/ healthcare resources consumption | 0-9 months
  iPCQ/iMCQ
Intervention costs | 0-9 months
  Cost analyses
Health status | 0-9 months
  EQ-5D-5L
Satisfaction with exercise intervention | 0-9 months
  Self-developed questionnaire
Biomarkers (systemic inflammation, growth factors, blood/brain barrier modulators) | 0-6 months
  Blood samples (plasma, serum, buffy coat and peripheral blood mononuclear cells (PBMC) )
Disease control | 0-9 months
  Progress or disease control of the breast cancer will be derived from medical records and/or the cancer registry
Cancer treatment | 0-9 months
  The type and duration of cancer treatment during the study will be derived from medical records and/or the cancer registry
Quality of working life | 0-9 months
  QWLQ-CS (add-on in several centers)

OTHER OUTCOMES:
Overall and breast-cancer specific survival | 0-60 months
  Exploratory outcome
Progression-free survival | 0-60 months
  Exploratory outcome
Safety of exercise intervention | 0-9 months
  (Serious) Adverse events potentially related to the exercise intervention
Urinary incontinence | 0-9 months
  Exploratory outcome (add on in some centers) - measured with ICIQ-UI
Maximal isokinetic and isometric leg strength, muscle thickness of m. rectus femoris (RF) and m. vastus lateralis (VL) | 0-9 months
  Exploratory outcome (add on in one center) - Isokinetic and isometric legstrength measured with peak torque / Muscle thickness with ultrasound protocol

CONTACTS AND LOCATIONS:
Overall Officials: Anne May, PhD, Principal Investigator — UMC Utrecht Julius Center
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kias A, Schmidt ME, Hiensch AE, Clauss D, Monninkhof EM, Pelaez M, Belloso J, Gunasekara N, Sweegers MG, Trevaskis M, Rundqvist H, Muller J, Wiskemann J, van der Wall E, Aaronson NK, Lachowicz M, Urruticoechea A, Zopf EM, Bloch W, Stuiver MM, Wengstrom Y, May AM, Steindorf K. Factors Associated With Employment and Quality of Working Life in Patients With Metastatic Breast Cancer. Cancer Med. 2025 Aug;14(15):e71074. doi: 10.1002/cam4.71074. PMID 40714912
- [Derived] Schouten AEM, Hiensch AE, Frederix GWJ, Monninkhof EM, Schmidt ME, Clauss D, Gunasekara N, Belloso J, Trevaskis M, Rundqvist H, Wiskemann J, Muller J, Sweegers MG, Fremd C, Altena R, Bijlsma RM, Sonke G, Lahuerta A, Mann GB, Francis PA, Richardson G, Malter W, Kufel-Grabowska J, van der Wall E, Aaronson NK, Senkus E, Urruticoechea A, Zopf EM, Bloch W, Stuiver MM, Wengstrom Y, Steindorf K, van der Meulen MP, May AM. Supervised Exercise for Patients With Metastatic Breast Cancer: A Cost-Utility Analysis Alongside the PREFERABLE-EFFECT Randomized Controlled Trial. J Clin Oncol. 2025 Apr 10;43(11):1325-1336. doi: 10.1200/JCO-24-01441. Epub 2025 Jan 13. PMID 39805062
- [Derived] Hiensch AE, Depenbusch J, Schmidt ME, Monninkhof EM, Pelaez M, Clauss D, Gunasekara N, Zimmer P, Belloso J, Trevaskis M, Rundqvist H, Wiskemann J, Muller J, Sweegers MG, Fremd C, Altena R, Gorecki M, Bijlsma R, van Leeuwen-Snoeks L, Ten Bokkel Huinink D, Sonke G, Lahuerta A, Mann GB, Francis PA, Richardson G, Malter W, van der Wall E, Aaronson NK, Senkus E, Urruticoechea A, Zopf EM, Bloch W, Stuiver MM, Wengstrom Y, Steindorf K, May AM. Supervised, structured and individualized exercise in metastatic breast cancer: a randomized controlled trial. Nat Med. 2024 Oct;30(10):2957-2966. doi: 10.1038/s41591-024-03143-y. Epub 2024 Jul 25. PMID 39054374
- [Derived] Pelaez M, Stuiver MM, Broekman M, Schmitz KH, Zopf EM, Clauss D, Wengstrom Y, Rosenberger F, Steindorf K, Urruticoechea A, May AM. Early Detection of Brain Metastases in a Supervised Exercise Program for Patients with Advanced Breast Cancer: A Case Report. Med Sci Sports Exerc. 2023 Oct 1;55(10):1745-1749. doi: 10.1249/MSS.0000000000003213. Epub 2023 May 12. PMID 37170950
- [Derived] Hiensch AE, Monninkhof EM, Schmidt ME, Zopf EM, Bolam KA, Aaronson NK, Belloso J, Bloch W, Clauss D, Depenbusch J, Lachowicz M, Pelaez M, Rundqvist H, Senkus E, Stuiver MM, Trevaskis M, Urruticoechea A, Rosenberger F, van der Wall E, de Wit GA, Zimmer P, Wengstrom Y, Steindorf K, May AM. Design of a multinational randomized controlled trial to assess the effects of structured and individualized exercise in patients with metastatic breast cancer on fatigue and quality of life: the EFFECT study. Trials. 2022 Jul 29;23(1):610. doi: 10.1186/s13063-022-06556-7. PMID 35906659
- See also: Website of the EFFECT study within the PREFERABLE project — https://www.h2020preferable.eu/
- See also: Twitter account PREFERABLE project — https://twitter.com/PREFERABLE_MBC